CLINICAL TRIAL: NCT05446766
Title: Feasibility Evaluation of a Self-guided Exposure-based Digital Intervention for Health Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Martin Kraepelien, Licensed clinical psychologist, Principal investigator, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEALTHANXIETY1
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Illness Anxiety Disorder; Somatic Symptom Disorder
Keywords: Self-guided intervention; Self-help; Digital intervention; Exposure therapy

STUDY DESIGN:
Masking Description: Psychological intervention, patient-reported outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-guided Exposure-based Digital Intervention for Health Anxiety (Experimental): Eight weeks of self-guided exposure-based intervention delivered digitally, via the Internet.
  Interventions: Behavioral: Self-guided Exposure-based Digital Intervention for Health Anxiety

INTERVENTIONS:
Behavioral: Self-guided Exposure-based Digital Intervention for Health Anxiety — An 8-week self-guided internet based CBT intervention which consists of text, exercises, examples and automated support. The format, potentially more accessible compared to traditional ICBT, will be developed with the aim to enhance treatment comprehension and motivation in the participants. The program consists of eight modules (chapters) where the main therapeutic focus is exposure with response prevention.
  Participant will be interviewed before the program starts, after 8 weeks and 3 months after the program ends. If in need for technical support, participant will be able to ask for assistance via the program and will then be contacted by a clinician via telephone within a couple of days.

SUMMARY:
This study investigates the feasibility and preliminary efficacy of a self-guided, exposure-based intervention for individuals who suffer from severe health anxiety. The study is a prospective single-group study based at Karolinska Institutet, Stockholm, Sweden, where 20-25 adults with DSM-5 Illness anxiety disorder or Somatic symptom disorder are enrolled in 8 weeks of unguided exposure-based treatment via the Internet. Outcomes include self-reported health anxiety symptoms, credibility and expectancy, adherence to the treatment protocol, client satisfaction, and negative events.

DETAILED DESCRIPTION:
Background

Severe health anxiety (Corresponding to a DSM-5-diagnosis of Illness anxiety disorder or somatic symptom disorder) is a condition associated with high distress, disability and increased health service utilization. Therapist guided Internet delivered cognitive behavioural therapy (ICBT) is efficacious in the treatment of severe health anxiety and has the advantage of requiring less treatment support per patient compared to traditional CBT, thus making the treatment more cost effective. Despite this, the access to ICBT is limited as it requires the active participation of a therapist. Given the relatively high prevalence of individuals experiencing excessive health anxiety, there is need for research on more accessible treatment options.

Unguided self-care interventions have the potential to improve access to treatment and increase cost-effectiveness and have a more immediate scalability. Also, unguided interventions have the advantage of being more easily disseminated outside the traditional mental health care systems and thus, have the potential to reach patients with subclinical, yet distressful, health anxiety.

Aim

The overall aim of this study is to develop a new internet-delivered CBT program based on exposure and response prevention - without therapist support - for patients with severe health anxiety and to examine its feasibility and potential clinical efficacy.

Design

This is a prospective single-group feasibility study with a pre-post design where a total of 25 participants with Illness anxiety disorder or Somatic symptom disorder (suffering from health anxiety) according to the Diagnostic and statistical manual of mental disorders 5 (DSM-5) are enrolled in an 8 weeks unguided internet based treatment targeting exposure and response prevention. The study will evaluate patient-reported satisfaction, engagement and adherence to treatment protocol, credibility, safety and pre-post changes in health anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A principal diagnosis Illness anxiety disorder or somatic symptom disorder (DSM-V)
* Access to a computer and the internet
* No serious medical illness
* Participants on psychotropic medication must have been on a stable dose for the last 4 weeks prior to baseline assessment

Exclusion Criteria:

* Difficulties to read or write that makes it hard to understand the content of the intervention
* Currently receiving similar psychological treatment for anxiety
* High risk of suicide
* Diagnosed with psychosis disorder or bipolar disorder
* Ongoing substance dependence
* Have an urgent need for more intensive psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Change in Health anxiety symptoms | pre-treatment assessment to 12 weeks after post-treatment assessment
  The Short health anxiety inventory - 14 item (SHAI-14). Higher scores indicate greater severity of health anxiety. Scores range from 0 to 42.
Adherence to the treatment: amount of exposures | Post-treatment assessment (immediately after treatment)
  Will be determined by the amount of exposure exercises reported in the program and in a weekly questionnaire. Acceptable level of adherence will be set to at least 50 % of participants working actively with exposure a majority of the days during a week for 4 weeks or more.
Adherence to the treatment: number of modules | Post-treatment assessment (immediately after treatment)
  Will be determined by the number of modules completed by the participants.
Adherence to the treatment: types of exposure | Post-treatment assessment (immediately after treatment)
  Will be determined by the number of different types of exposure exercises performed by participants. At the end of the program, participants will answer yes or no to whether they engaged in each component (type of exposure exercise) of the intervention.
Unintended treatment effects | Post-treatment assessment (immediately after treatment)
  Participants will be asked to state whether they had experienced any negative or unwanted effects of the treatment. If answering 'Yes', participants will be asked to specify the adverse event in free text. Adverse events will primarily be reported as the total number of reported events.
Satisfaction with treatment | Post-treatment assessment (immediately after treatment)
  Client Satisfaction Questionnaire (CSQ-8). Scores range from 8-32 with higher scores indicating greater satisfaction. An average Client Satisfaction Questionnaire-8 score of at least 22 will provide support for the acceptability and feasibility of this intervention.

SECONDARY OUTCOMES:
Change in Health anxiety symptoms | pre-treatment assessment to Post-treatment assessment (immediately after treatment)
  The Short health anxiety inventory - 14 item (SHAI-14). Higher scores indicate greater severity of health anxiety. Scores range from 0 to 42.
Change in Health anxiety symptoms | pre-treatment assessment to 4 weeks after post-treatment assessment
  The Short health anxiety inventory - 14 item (SHAI-14). Higher scores indicate greater severity of health anxiety. Scores range from 0 to 42.
Change in depressive symptoms | pre-treatment assessment to12 weeks after post-treatment assessment
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27.
Change in depressive symptoms | pre-treatment assessment to Post-treatment assessment (immediately after treatment)
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27.
Change in depressive symptoms | pre-treatment assessment to 4 weeks after post-treatment assessment
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27.
Change in diagnostic status | Change from baseline interview to 12 weeks after post-treatment assessment
  Health Preoccupation Diagnostic Interview (HPDI). HPDI is a structured interview designed to assess Illness anxiety disorder and Somatic symptom disorder according to DSM-V criteria. HPDI will be administered via telephone.
Change in anxiety symptoms | pre-treatment assessment to 12 weeks after post-treatment assessment
  Generalized Anxiety Disorder 7-item scale (GAD-7). Higher total scores indicate greater severity of anxiety symptoms. Scores range from 0 to 21.
Change in anxiety symptoms | pre-treatment assessment to Post-treatment assessment (immediately after treatment)
  Generalized Anxiety Disorder 7-item scale (GAD-7). Higher total scores indicate greater severity of anxiety symptoms. Scores range from 0 to 21.
Change in anxiety symptoms | pre-treatment assessment to 4 weeks after post-treatment assessment
  Generalized Anxiety Disorder 7-item scale (GAD-7). Higher total scores indicate greater severity of anxiety symptoms. Scores range from 0 to 21.
Change in life quality | pre-treatment assessment to 12 weeks after post-treatment assessment
  Brunnsviken Brief Quality of Life Questionnaire (BBQ). A 12-item questionnaire covering six different life domains: leisure time, view on life, creativity, learning, friends and friendship, and view of self. Scores range from 0 to 96, where higher values indicate higher quality of life satisfaction.
Change in life quality | pre-treatment assessment to Post-treatment assessment (immediately after treatment)
  Brunnsviken Brief Quality of Life Questionnaire (BBQ). A 12-item questionnaire covering six different life domains: leisure time, view on life, creativity, learning, friends and friendship, and view of self. Scores range from 0 to 96, where higher values indicate higher quality of life satisfaction.
Credibility/expectancy | week 3 of treatment
  The five-item version of Credibility/Expectancy Questionnaire (CEQ). The CEQ ranges from 0 to 10 points per item and 0 to 50 points in total, where a higher score reflects better treatment credibility.
Usability | Post-treatment assessment (immediately after treatment)
  The System Usability Scale (SUS). The SUS consists of ten items, with a range of 0-4 points per item. The items are summed up and calculated with a formula resulting in a total score between 0 and 100, with a higher score reflecting better system usability.
Experience with the program | Post-treatment assessment (immediately after treatment)
  A non-validated questionnaire measuring experience working with the program. The scale comprises four questions where participant answer whether the intervention was perceived as likable, easy to understand, whether examples given felt relevant and whether functionality and information contributed to the participant feeling overwhelmed. Answers will be made on a four-point scale ranging from 0 (strongly disagree) to 3 (strongly agree). It will be optional to add a free-text comment to the responses, as well as suggestions of overall improvements.
Post-treatment adherence to exposure exercises | 12 weeks after post-treatment assessment
  Adherence to the exposure exercises will be determined by an online questionnaire where participant on a four point Likert scale will state to what extent they have worked with exposure: "not at all", "occasionally", "more than half of the days" and "daily".

OTHER OUTCOMES:
Telephone interview | immediately after treatment
  A semi-structured interview concerning the experience of the intervention and format will be conducted via telephone

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum för Psykiatriforskning, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual data will be available upon reasonable request.

REFERENCES:
- [Derived] Osterman S, Hentati A, Forsell E, Axelsson E, Hedman-Lagerlof E, Lindefors N, Ivanov VZ, Kraepelien M. Brief digital self-care intervention for health anxiety in a Swedish Medical University Clinic: a prospective single-group feasibility study. BMJ Open. 2023 Dec 21;13(12):e077376. doi: 10.1136/bmjopen-2023-077376. PMID 38135329